CLINICAL TRIAL: NCT04246489
Title: A Phase II, Multicenter, Open Label Study of Bintrafusp Alfa (M7824) Monotherapy in Participants With Advanced, Unresectable Cervical Cancer With Disease Progression During or After Platinum-Containing Chemotherapy
Brief Title: Bintrafusp Alfa Monotherapy in Platinum-Experienced Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS200647_0017; 2019-003583-40 (EudraCT Number)
Record Dates: First submitted 2020-01-28; First posted 2020-01-29 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Uterine Cervical Neoplasms
Keywords: M7824; INTR@PID; Bintrafusp alfa; programmed death-ligand 1; Cervical Cancer; Transforming growth factor-β (TGF-β)
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bintrafusp alfa (Experimental)
  Interventions: Drug: Bintrafusp alfa

INTERVENTIONS:
Drug: Bintrafusp alfa — Participants received an intravenous infusion of 1200 milligrams (mg) bintrafusp alfa once every 2 weeks until confirmed disease progression, death, unacceptable toxicity and study withdrawal.
  Other Names: M7824

SUMMARY:
The main purpose of this study was to evaluate clinical efficacy and safety of bintrafusp alfa in participants with advanced, unresectable cervical cancer with disease progression during or after platinum-containing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants who had advanced unresectable and/or metastatic cervical cancer (squamous cell carcinoma, adenocarcinoma, adenosquamous cell carcinoma) with disease progression during or after the prior platinum-containing chemotherapy:

  1. The prior platinum-containing chemotherapy may be a systemic treatment for advanced unresectable, recurrent, persistent or metastatic disease or treatment in the adjuvant or neo-adjuvant setting with disease progression or recurrence within 6 months of completion of platinum-containing chemotherapy
  2. Participants who previously only received platinum as a radiosensitizer are not eligible
  3. Participants must be naïve to checkpoint inhibitors
* Participants who had measurable disease
* Participants who provide a tumor tissue sample, either from archival tissue or newly obtained core or excisional biopsy. If the participant received local therapy (For example: radiation therapy or chemoradiotherapy) after the archival tissue was taken, a new biopsy was required
* Participants who had Eastern Cooperative Oncology Group (ECOG) PS of 0 to 1
* Life expectancy greater than or equals to (>=) 12 weeks as judged by the Investigator
* Adequate hematological, hepatic and renal function as defined in the protocol
* Participants with known Human Immunodeficiency Virus (HIV) infections were in general eligible if the following criteria are met:

  1. Clinically indicated participants must be stable on antiretroviral therapy (ART) for at least 4 weeks and agree to adhere to ART
  2. had no evidence of documented multi-drug resistance that would prevent effective ART
  3. had an HIV viral load of < 400 copies per milliliter (/mL) at Screening
  4. had CD4+ T-cell (CD4+) counts >= 350 cells/microliter
  5. For participants with a history of an Acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within the last 12 months, participants may be eligible only after consultation and agreement with the study Medical Monitor
  6. If prophylactic antimicrobial drugs were indicated, participants would still be considered eligible upon agreement with the study Medical Monitor
* Participants with hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infections were in general eligible if the following criteria are met:

  1. HBV viral load below the limit of quantification. If medically indicated, participants infected with HBV must be treated and on a stable dose of antivirals at study entry and with planned monitoring and management according to appropriate labeling guidance
  2. Participants with a history of HCV infection should have completed curative antiviral treatment and require HCV viral load below the limit of quantification
  3. Participants on concurrent HCV treatment should have HCV below the limit of quantification
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with active central nervous system (CNS) metastases causing clinical symptoms or require therapeutic intervention are excluded. Participants with a history of treated CNS metastases (by surgery or radiation therapy) are not eligible unless they have fully recovered from treatment, demonstrated no progression for at least 4 weeks, and are not using steroids for at least 7 days prior to the start of study treatment
* Participants with interstitial lung disease or has had a history of pneumonitis that has required oral or intravenous (IV) steroids
* Participants with significant acute or chronic infections
* Participants with active autoimmune disease that might deteriorate when receiving an immunostimulatory agent
* Participants with clinically significant cardiovascular/cerebrovascular disease including: cerebral vascular accident/stroke, myocardial infarction, unstable angina, congestive heart failure, or serious cardiac arrhythmia
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (73):
- United States (11):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - Stanford University Hospital and Clinics - Stanford Cancer Center, Stanford, California
  - The Stamford Hospital, Stamford, Connecticut
  - Karmanos Cancer Institute, Farmington Hills, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - UC Health Clinical Trials Office, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The West Clinic, Germantown, Tennessee
  - SCRI - Tennessee Oncology, Nashville, Tennessee
- Argentina (3):
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Sanatorio El Parque, Salta
  - Centro Medico San Roque S.R.L., San Miguel de Tucumán
- Australia (3):
  - Peter MacCallum Cancer Centre-East Melbourne, Melbourne
  - Linear Clinical Research Limited, Nedlands
  - Calvary Mater Newcastle, Waratah
- Belgium (8):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Gent - Pneumology, Ghent
  - AZ Groeninge - Campus Kennedylaan - account 2, Kortrijk
  - CHU de Liège - PARENT, Liège
  - CHU Sart Tilman, Liège
  - UZ Leuven, Pellenberg
  - GZA Ziekenhuizen - Campus Sint-Augustinus, Wilrijk
- Brazil (3):
  - HGB - Hospital Giovanni Battista - Mãe de Deus Center - Centro de Pesquisa Clínica - Instituto do Câncer, Porto Alegre
  - Clínica de Pesquisas e Centro de Estudos em Oncologia Ginecológica e Mamária Ltda., São Paulo
  - IBCC - Instituto Brasileiro de Controle do Câncer, São Paulo
- China (7):
  - Chongqing Cancer Hospital, Chongqing
  - Sun Yat-sen University, Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - Shanghai Cancer Hospital, Fudan University, Shanghai
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital, Zhengzhou
- France (10):
  - Institut Bergonié, Bordeaux
  - Centre Oscar lambret - Service d'Oncologie medicale, Lille
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hôpital Cochin - Hematologie et Oncologie Médicale, Paris
  - Centre Hospitalier Lyon Sud - service d'oncologie medicale, Pierre-Bénite
  - CARIO - Centre Armoricain de Radiothérapie, Imagerie médicale et Oncologie, Plérin
  - Institut Jean Godinot - Service d'hématologie et Oncologie Médicale, Reims
  - ICO - Site René Gauducheau, Saint-Herblain
  - Institut de Cancérologie de Strasbourg Europe - ICANS - Service d'oncologie médicale, Strasbourg
- Hungary (2):
  - Orszagos Onkologiai Intezet - Nogyogyaszati Osztaly, Budapest
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz - Onkoradiologia, Nyíregyháza
- Japan (10):
  - National Cancer Center Hospital - Dept of Mammary Gland/Oncology, Chūōku
  - NHO Kyushu Cancer Center - Dept of Gynecology, Fukuoka
  - Saitama Medical University International Medical Center - Dept of Gynecology/Oncology, Hidaka-shi
  - Cancer Institute Hospital of JFCR - Dept of Gynecology, Kōtoku
  - Kurume University Hospital - Dept of Gynecology, Kurume-shi
  - Jikei University Hospital - Dept of Gynecology, Minatoku
  - University Hospital, University of the Ryukyus - Dept of Obstetrics/Gynecology, Nakagami-gun
  - Osaka International Cancer Institute - Dept of Gynecology, Osaka
  - NHO Hokkaido Cancer Center - Dept of Gynecology, Sapporo
  - Kanagawa Cancer Center - Dept of Gynecology, Yokohama
- Russia (2):
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
  - LLC "ClinicaUZI4D", Pyatigorsk
- South Korea (6):
  - National Cancer Center, Goyang-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Ajou University Hospital, Suwon
- Spain (8):
  - Hospital Clinic i Provincial de Barcelona - Servicio de Oncologia, Barcelona
  - Hospital Universitari Vall d'Hebron - Dept of Oncology, Barcelona
  - ICO Girona - Hospital Doctor Josep Trueta - Servicio de Oncologia Medica, Girona
  - Clinica Universidad de Navarra (MAD) - Oncology Service, Madrid
  - Hospital Universitario 12 de Octubre - Servicio de Oncologia, Madrid
  - Hospital Universitario Ramon y Cajal - Servicio de Oncologia, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Clinico Universitario de Valencia - Servicio de Hematologia y Oncologia Medica, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, EMD Serono will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.emdgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Background] Strauss J, Heery CR, Schlom J, Madan RA, Cao L, Kang Z, Lamping E, Marte JL, Donahue RN, Grenga I, Cordes L, Christensen O, Mahnke L, Helwig C, Gulley JL. Phase I Trial of M7824 (MSB0011359C), a Bifunctional Fusion Protein Targeting PD-L1 and TGFbeta, in Advanced Solid Tumors. Clin Cancer Res. 2018 Mar 15;24(6):1287-1295. doi: 10.1158/1078-0432.CCR-17-2653. Epub 2018 Jan 3. PMID 29298798
- [Background] Lan Y, Zhang D, Xu C, Hance KW, Marelli B, Qi J, Yu H, Qin G, Sircar A, Hernandez VM, Jenkins MH, Fontana RE, Deshpande A, Locke G, Sabzevari H, Radvanyi L, Lo KM. Enhanced preclinical antitumor activity of M7824, a bifunctional fusion protein simultaneously targeting PD-L1 and TGF-beta. Sci Transl Med. 2018 Jan 17;10(424):eaan5488. doi: 10.1126/scitranslmed.aan5488. PMID 29343622
- [Background] Vugmeyster Y, Grisic AM, Wilkins JJ, Loos AH, Hallwachs R, Osada M, Venkatakrishnan K, Khandelwal A. Model-informed approach for risk management of bleeding toxicities for bintrafusp alfa, a bifunctional fusion protein targeting TGF-beta and PD-L1. Cancer Chemother Pharmacol. 2022 Oct;90(4):369-379. doi: 10.1007/s00280-022-04468-6. Epub 2022 Sep 6. PMID 36066618
- [Derived] Birrer M, Li G, Yunokawa M, Lee JY, Kim BG, Oppermann CP, Zhou Q, Nishio S, Okamoto A, Wu X, Mileshkin L, Oaknin A, Ray-Coquard I, Hasegawa K, Jehl G, Vugmeyster Y, Zhang S, Bajars M, Yonemori K. Bintrafusp Alfa for Recurrent or Metastatic Cervical Cancer After Platinum Failure: A Nonrandomized Controlled Trial. JAMA Oncol. 2024 Sep 1;10(9):1204-1211. doi: 10.1001/jamaoncol.2024.2145. PMID 39052242
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200647_0017
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 203 participants were screened, of which 146 participants received bintrafusp alfa monotherapy.
Groups:
- Bintrafusp Alfa: Participants received an intravenous infusion of 1200 milligrams (mg) bintrafusp alfa once every 2 weeks until confirmed disease progression, unacceptable toxicity, study withdrawal or death.
Period: Overall Study
Arm/Group | Bintrafusp Alfa
Started | 146
Completed | 146
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) included all participants, who were administered at least one dose of bintrafusp alfa.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 132
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 90
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 37
  More than one race | 0
  Unknown or Not Reported | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC)
Description: Confirmed objective response was defined as the number of participants with a confirmed objective response of complete response (CR) or partial response (PR). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Confirmed CR = at least 2 determinations of CR at least 4 weeks apart and before progression. Confirmed PR = at least 2 determinations of PR at least 4 weeks apart and before progression (and not qualifying for a CR). Confirmed objective response was determined according to RECIST v1.1 and as adjudicated by IRC.
Time Frame: Time from first treatment up to 688 days
Population: FAS included all participants who were administered at least one dose of bintrafusp alfa.
Measure: Count of Participants; unit: Participants
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 146
Participants | 32

2. Secondary Outcome: Duration of Response (DOR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC)
Description: DOR was defined for participants with confirmed response, as the time from first documentation of confirmed objective response (Complete Response [CR] or Partial Response [PR]) according to RECIST 1.1 to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DOR was determined according to RECIST v1.1 and assessed by IRC. Results were calculated based on Kaplan-Meier estimates.
Time Frame: Time from first treatment up to 688 days
Population: FAS included all participants who were administered at least one dose of bintrafusp alfa.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 146
months | NA [7.4 to NA] — The median was not reached, and the upper limit could not be estimated due to insufficient number of events

3. Secondary Outcome: Durable Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC)
Description: Durable Response was defined as the number of participants with confirmed objective response (CR or PR) according to RECIST 1.1, determined by IRC with duration of at least 6 months. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from first treatment up to 688 days
Population: FAS included all participants who were administered at least one dose of bintrafusp alfa.
Measure: Count of Participants; unit: Participants
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 146
Participants | 19

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related TEAEs, Including Adverse Event of Special Interests (AESIs)
Description: Adverse Event (AE) was defined any untoward medical occurrence in a participant administered with a study drug, which does not necessarily had a causal relationship with this treatment. Serious AE was defined AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs: TEAEs was defined as events with onset date or worsening during the on-treatment period. TEAEs included serious AEs and non-serious AEs. Treatment-related TEAEs: reasonably related to the study intervention. AESIs included Infusion-related reactions, Immune-related AEs, Transforming growth factor- beta (TGF-ß) inhibition mediated skin AE, bleeding and anemia.
Time Frame: Time from first treatment up to 688 days
Population: Safety analysis set included all participants who were administered at least one dose of bintrafusp alfa
Measure: Count of Participants; unit: Participants
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 146
Participants
  TEAE's | 145
  Treatment Related TEAEs | 106
  AESI: Infusion-related reaction | 5
  AESI: Immune-related AE | 49
  AESI: TGF-beta inhibition mediated skin AE | 7
  AESI: Anemia | 82
  AESI: Bleeding events | 81

5. Secondary Outcome: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) Assessed by Independent Review Committee (IRC)
Description: PFS was defined as the time from first administration of study intervention until date of the first documentation of disease progression (PD) or death due to any cause, whichever occurred first. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. Kaplan-Meier estimates was used to calculate PFS.
Time Frame: Time from first administration of study drug until the first documentation of PD or death, assessed up to 688 days
Population: FAS included all participants who were administered at least one dose of bintrafusp alfa.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 146
months | 1.9 [1.8 to 2.2]

6. Secondary Outcome: Number of Participants With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by the Investigator
Description: Confirmed objective response was defined as the number of participants with a confirmed objective response of complete response (CR) or partial response (PR). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Confirmed CR = at least 2 determinations of CR at least 4 weeks apart and before progression. Confirmed PR = at least 2 determinations of PR at least 4 weeks apart and before progression (and not qualifying for a CR). Confirmed objective response was determined according to RECIST v1.1 and as adjudicated by Investigator.
Time Frame: Time from first treatment up to 688 days
Population: FAS included all participants who were administered at least one dose of bintrafusp alfa.
Measure: Count of Participants; unit: Participants
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 146
Participants | 25

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first administration of study intervention to the date of death due to any cause. The OS was analyzed by using the Kaplan-Meier method.
Time Frame: Time from first administration of study drug up to data cutoff (assessed up to 688 days)
Population: FAS included all participants who were administered at least one dose of bintrafusp alfa.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 146
months | 13.7 [10.6 to 17.1]

8. Secondary Outcome: Serum Pre-Dose Concentrations (Ctrough) of Bintrafusp Alfa
Description: Ctrough was defined as the concentration observed immediately before next dosing (corresponding to pre-dose or trough concentration for multiple dosing).
Time Frame: At Day 15, Day 29, Day 43, Day 85, Day 127, Day 169, Day 253, Day 337, Day 421, Day 505 and Day 589
Population: Pharmacokinetic (PK) analysis set included all participants who completed at least one dose of bintrafusp alfa and who provided at least one sample with a measurable concentration of bintrafusp alfa. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at specified time points for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 143
microgram per milliliter (mcg/mL)
  Day 15: number analyzed (Participants) | 125
  Day 15 | 73.7 (55.3)
  Day 29: number analyzed (Participants) | 103
  Day 29 | 107 (48.7)
  Day 43: number analyzed (Participants) | 84
  Day 43 | 108 (53)
  Day 85: number analyzed (Participants) | 47
  Day 85 | 115 (44.9)
  Day 127: number analyzed (Participants) | 35
  Day 127 | 107 (69)
  Day 169: number analyzed (Participants) | 25
  Day 169 | 137 (41)
  Day 253: number analyzed (Participants) | 12
  Day 253 | 101 (45.8)
  Day 337: number analyzed (Participants) | 11
  Day 337 | 120 (50.9)
  Day 421: number analyzed (Participants) | 5
  Day 421 | 103 (56.4)
  Day 505: number analyzed (Participants) | 4
  Day 505 | 220 (22.4)
  Day 589: number analyzed (Participants) | 3
  Day 589 | 154 (10.4)

9. Secondary Outcome: Serum Concentration at End of Infusion (CEOI) of Bintrafusp Alfa
Description: Serum Concentration at End of Infusion (CEOI) of bintrafusp alfa is reported.
Time Frame: At Day 1 and Day 29
Population: PK analysis set included all participants who completed at least one dose of Bintrafusp Alfa and who provided at least one sample with a measurable concentration of Bintrafusp Alfa. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at specified time points for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 143
mcg/mL
  Day 1: number analyzed (Participants) | 142
  Day 1 | 469 (21.9)
  Day 29: number analyzed (Participants) | 102
  Day 29 | 546 (24.1)

10. Secondary Outcome: Number of Participants With Positive Antidrug Antibodies (ADA)
Description: Serum samples were analyzed by a validated assay method to detect the presence of antidrug antibodies (ADA). Number of participants with positive ADA were reported.
Time Frame: Time from first treatment up to 688 days
Population: Immunogenicity analysis set included all participants who received at least one dose of bintrafusp alfa and who had at least one valid result of ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 142
Participants | 33

11. Secondary Outcome: Percentage of Participants With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC) According to Programmed Death Ligand 1 (PD-L1) Expression
Description: Confirmed objective response was defined as the percentage of participants with a confirmed objective response of complete response (CR) or partial response (PR). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Confirmed CR = at least 2 determinations of CR at least 4 weeks apart and before progression. Confirmed PR = at least 2 determinations of PR at least 4 weeks apart and before progression (and not qualifying for a CR). Confirmed objective response was determined according to RECIST v1.1 and as adjudicated by IRC through PD-L1 Subgroup. Participants with PD-L1 positive tumors (Combined positive score (CPS) >=1) and PD-L1 negative tumors (CPS<1).
Time Frame: Time from first treatment up to 688 days
Population: FAS included all participants who were administered at least one dose of bintrafusp alfa. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at specified categories for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 141
percentage of participants
  PD-L1 positive tumors (CPS>=1): number analyzed (Participants) | 86
  PD-L1 positive tumors (CPS>=1) | 25.6 [16.8 to 36.1]
  PD-L1 negative tumors (CPS <1): number analyzed (Participants) | 55
  PD-L1 negative tumors (CPS <1) | 18.2 [9.1 to 30.9]

12. Secondary Outcome: PFS According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC) According to Programmed Death Ligand 1 (PD-L1) Expression
Description: PFS was defined as the time from first administration of study intervention until the first documentation of disease progression (PD) or death due to any cause, whichever occurred first. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. PFS was determined according to RECIST v1.1 and as adjudicated by IRC through PD-L1 Subgroup. Participants with PD-L1 positive tumors (Combined positive score (CPS) >=1) and PD-L1 negative tumors (CPS<1).
Time Frame: Time from first administration of study drug until the first documentation of PD or death, assessed up to 688 days
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 141
months
  PD-L1 positive tumors (CPS>=1): number analyzed (Participants) | 86
  PD-L1 positive tumors (CPS>=1) | 1.9 [1.8 to 4.3]
  PD-L1 negative tumors (CPS<1): number analyzed (Participants) | 55
  PD-L1 negative tumors (CPS<1) | 1.9 [1.7 to 2.0]

13. Secondary Outcome: Overall Survival (OS) as Assessed According to Programmed Death Ligand 1 (PD-L1) Expression
Description: OS was defined as the time from first administration of study intervention to the date of death due to any cause. The OS was analyzed by using the Kaplan-Meier method. Participants with PD-L1 positive tumors (Combined positive score (CPS) >=1) and PD-L1 negative tumors (CPS<1).
Time Frame: Time from first administration of study drug up to 688 days
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 141
months
  PD-L1 positive tumors (CPS>=1): number analyzed (Participants) | 86
  PD-L1 positive tumors (CPS>=1) | 17.5 [12.5 to NA] — Due to small number of events Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derived.
  PD-L1 negative tumors (CPS<1): number analyzed (Participants) | 55
  PD-L1 negative tumors (CPS<1) | 8.7 [5.8 to 11.8]

ADVERSE EVENTS:
Time Frame: Time from first treatment up to 688 days
Arm/Group | Bintrafusp Alfa
All-Cause Mortality (participants affected / at risk) | 76/146
Serious Adverse Events (participants affected / at risk) | 94/146
Other Adverse Events (participants affected / at risk) | 139/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bintrafusp Alfa (N=146)
Anaemia (Blood and lymphatic system disorders) | 14
Blood loss anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Immune-mediated thyroiditis (Endocrine disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Secondary adrenocortical insufficiency (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Anal haemorrhage (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 4
Dental caries (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Obstructive defaecation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Disease progression (General disorders) | 12
General physical health deterioration (General disorders) | 4
Malaise (General disorders) | 1
Pain (General disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Hepatic pain (Hepatobiliary disorders) | 1
Abdominal sepsis (Infections and infestations) | 1
Brain abscess (Infections and infestations) | 1
Intestinal fistula infection (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic arthritis streptococcal (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Urinary tract infection bacterial (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Radiation proctitis (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Stoma obstruction (Injury, poisoning and procedural complications) | 1
Amylase increased (Investigations) | 1
Lipase increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2
Malnutrition (Metabolism and nutrition disorders) | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 2
Brain oedema (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Myasthenia gravis (Nervous system disorders) | 1
Neuritis (Nervous system disorders) | 1
Polyneuropathy in malignant disease (Nervous system disorders) | 1
Device dislocation (Product Issues) | 2
Acute kidney injury (Renal and urinary disorders) | 3
Cystitis haemorrhagic (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 15
Haemorrhage urinary tract (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 3
Renal failure (Renal and urinary disorders) | 2
Ureteral polyp (Renal and urinary disorders) | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Female genital tract fistula (Reproductive system and breast disorders) | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bintrafusp Alfa (N=146)
Anaemia (Blood and lymphatic system disorders) | 80
Hyperthyroidism (Endocrine disorders) | 10
Hypothyroidism (Endocrine disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 22
Diarrhoea (Gastrointestinal disorders) | 12
Gingival bleeding (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 30
Stomatitis (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 20
Asthenia (General disorders) | 23
Oedema peripheral (General disorders) | 12
Pyrexia (General disorders) | 25
Urinary tract infection (Infections and infestations) | 14
Alanine aminotransferase increased (Investigations) | 20
Amylase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 19
Blood alkaline phosphatase increased (Investigations) | 10
Blood creatinine increased (Investigations) | 9
Lipase increased (Investigations) | 10
Weight decreased (Investigations) | 8
Decreased appetite (Metabolism and nutrition disorders) | 24
Hypoalbuminaemia (Metabolism and nutrition disorders) | 15
Hypokalaemia (Metabolism and nutrition disorders) | 12
Hyponatraemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 10
Headache (Nervous system disorders) | 11
Insomnia (Psychiatric disorders) | 11
Haematuria (Renal and urinary disorders) | 26
Vaginal haemorrhage (Reproductive system and breast disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 17
Rash (Skin and subcutaneous tissue disorders) | 24
Fatigue (General disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT04246489/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT04246489/SAP_001.pdf